CLINICAL TRIAL: NCT03733548
Title: Improving Emotion Regulation in Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20013904
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Adhd
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Pilot trial to finish developing and refining the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regulating Emotions Like An eXpert (RELAX) (Experimental): Families at the Virginia Commonwealth University Center for Psychological Services and Development or Clark-Hill Institute for Positive Youth Development
  Interventions: Behavioral: RELAX

INTERVENTIONS:
Behavioral: RELAX — Regulating Emotions Like An eXpert (RELAX) consists of 8 weekly, 90-minute sessions delivered (60 minutes of parents and adolescents meeting separately, 30 minutes of a combined meeting) in a group format. RELAX equips adolescents with emotion regulation and conflict management skills. This program includes a parent involvement component designed to help parents support adolescents' use of these skills. Each week skills will be discussed and practiced in group, and a skills rehearsal homework activity will be assigned. Following the program, an 8-week follow-up review session will be offered. Additionally, a single 60 minute focus group will be held following the review session to solicit parent and adolescent feedback on the intervention.

SUMMARY:
The purpose of our study is to examine the impact of a program that provides emotion regulation skills for adolescents aged 11-16 with Attention-Deficit/Hyperactivity Disorder (ADHD) and poor emotion regulation. The program is called RELAX (Regulating Emotions Like An eXpert). RELAX is an experimental intervention that may equip adolescents with emotion regulation and conflict management skills and includes parent involvement to help parents support adolescents' use of these skills.

DETAILED DESCRIPTION:
Regulating Emotions Like An eXpert (RELAX) consists of 8 weekly 90-minute group sessions and 1 booster session 8 weeks after the completion of the RELAX intervention. The first 60 minutes of each group involve separate parent and adolescent groups. Adolescents (ages 11-16) attend an emotion regulation and conflict management skills group, while parents attend a group focused on how to support utilization of these skills in adolescents at home and school through use of modeling their own emotion regulation skills and use of supportive emotion socialization practices. For the final 30 minutes of the session, parents and adolescents combine and complete a collaborative activity and skill rehearsal homework is discussed for the week. Homework will be discussed at the beginning of the separate group meetings the following week. The primary overall goal of the RELAX intervention is to assist adolescents and parents in traveling down the Path of RELAXation by working on the three C's (communication, coping, and conflict management skills). A multimethod assessment of emotional, social, and family functioning will be assessed pre- and post-intervention and at an 8 week follow-up.

ELIGIBILITY:
Inclusion Criteria (adolescents):

* ADHD diagnosis
* parent-reported emotion regulation in the clinical range
* full scale intelligence quotient ≥80
* English as a primary language

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Emotion Dysregulation | Baseline, Post-Intervention (Completion of 8 week intervention), 8 week Follow-up (Approximately 2 months after completion of intervention)
  Parent and adolescent-reported emotion regulation on the Difficulties in Emotion Regulation Scale (DERS; Bunford et al., 2018; Kaufman et al., 2016). Total score is out of 180 (5 point Likert for each of 36 items). Higher scores indicate more difficulties with emotion regulation. RSA will be assessed with an EKG: three electrodes will be placed in a bipolar configuration on the left and right rib cage and the sternum. RSA is a measure of heart rate variability based on the respiratory cycle and is an indicator of vagal regulation (Berntson, Cacioppo, & Quigley, 1997). Decreases in RSA, or RSA withdrawal, correspond to increased heart-rate and arousal; whereas, increases in RSA, or RSA augmentation, correspond to decreased arousal.
Change in Family Conflict | Baseline, Post-Intervention (Completion of 8 week intervention), 8 week Follow-up (Approximately 2 months after completion of intervention)
  Parent and adolescent-reported family conflict as measured by the Conflict Behavior Questionnaire (CBQ). The CBQ consists of 20 true-false questions, with higher scores indicating more conflict between parents and their children.

SECONDARY OUTCOMES:
Emotion Reactivity Predicting Treatment Outcomes | Baseline, Post-Intervention (Completion of 8 week intervention), 8 week Follow-up (Approximately 2 months after completion of intervention)
  Baseline respiratory sinus arrhythmia (RSA) and RSA-Reactivity Predicting Change in Emotion Regulation and Family Conflict.
Change in Emotion Socialization Predicting Treatment Outcomes | Baseline, Post-Intervention (Completion of 8 week intervention)
  Observed emotion socialization predicting Emotion Regulation and Family Conflict. Observational emotion socialization will be coded during a parent-adolescent conflict discussion task. During this task adolescents will be instructed to share a recent parent-adolescent conflict that was a stressor for them, and the dyad will discuss the recent conflict for five minutes. The discussions will be coded for parent responses to adolescents' distress through seven possible reactions: emotion-focused, problem-focused, minimizing, punitive; magnifying, autonomy-inhibiting, and facilitative engagement. Responses will be coded on a 4-point scale representing an (1) absence, (2) minimal, (3) moderate, or (4) strong presence of the behavior reflected in each of the codes.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Langberg, PhD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Clark-Hill Institute for Positive Youth Development, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.